CLINICAL TRIAL: NCT04771702
Title: Propofol Measurement in Expiration Air and Monitoring of EEG and Pain in Patients Undergoing Low Back Surgery
Brief Title: Expired Propofol in Low Back Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Johan C Ræder, Professor, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Edmon-Oslo-Low Back Surgery
Record Dates: First submitted 2021-01-13; First posted 2021-02-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Anesthesia

STUDY DESIGN:
Intervention Model Description: The intervention is to have patients in 20 min stable anaesthesia before start of surgery in order to validate the use of exhaled propofol versus pharmakokinetic modelling and measured plasma concentration
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Edmon arm (Experimental)
  Interventions: Device: Edmon

INTERVENTIONS:
Device: Edmon — Exhaled air will be analyzed for propofol

SUMMARY:
Edmon (BBraun, Germany) is a portable, commercially available device for measurement of propofol in exhaled air.

The study will aim at evaluating the sensitivity and specificity of such exhaled propofol values compared with plasma propofol and measures of anaesthetic and antinociceptive effect.

DETAILED DESCRIPTION:
Elective low-back surgery patients will be induced for general intubation anesthesia with propofol and remifentanil.

After induction a 20 min period of stable propofol infusion only will be established before start of surgery. The patients will be monitored for exhaled propofol, plasma propofol (blood samples), continous frontal EEG, Bispectral Index (BIS), skin conductance, estimated (computer based) concentrations of plasma and effect site propofol, and skin conductance.

After start of surgery (with ongoing propofol and restart of remifentanil TCI) the monitoring will continue in order to explore these relationships further.

ELIGIBILITY:
Inclusion Criteria:

* Elective patients scheduled for low-back surgery
* BMI between 20 -32 kg/m2
* ASA I-II
* Written informed concent

Exclusion Criteria:

* Contraindication to propofol TCI
* Use of psychopharmaco or neurologic disease
* Pregnancy or breast feeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Exhaled air versus plasma concentration | per-operative

SECONDARY OUTCOMES:
EEG recording | per-operative
  EEG will be recorded and compared with plasma propofol, exhaled propofol and BIS
Exhaled propofol 2 | per-operative
  Exhaled propofol versus dose given, estimated plasma concentration, estimated effect site concentration
Nociceptive stimulation | per-operative
  Skin conductance versus plasma and exhaled propofol concentration

CONTACTS AND LOCATIONS:
Overall Officials: Kristin S Thagaard, MD, Study Director — Oslo University Hospital
Locations (1):
- Dept of Anesthesiology, Oslo University Hospital, Ullevaal, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No